CLINICAL TRIAL: NCT05983718
Title: Comparison of Positional Accuracy in Dental Implant Placement Between Conventionally Used Guide Pin and 3D Printed Surgical Guide Developed From CBCT
Brief Title: A Study of Surgical Guide Assisted Dental Implantation in Bangladesh
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dhaka Dental College and Hospital (Other)
Collaborators: Bangladesh University of Engineering and Technology (Other)
Responsible Party: Principal Investigator, Dr. Md. Al-Amin Sarkar, Junior Consultant, Dhaka Dental College and Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BME-BUET-DDCH-001
Record Dates: First submitted 2023-08-02; First posted 2023-08-09 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Partially Edentulous Mandible; Dental Implantation

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FREE HAND (GUIDE-PIN-assisted) (Active Comparator)
  Interventions: Procedure: Guide-pin-assisted Freehand surgery
- FULL GUIDED (Experimental)
  Interventions: Device: Surgical Guide

INTERVENTIONS:
Device: Surgical Guide — For this case, after the patient is given anesthesia, the guide will be placed on the teeth. All the drillings will be performed through the guided path. There will be no need for raising flap according to flapless surgery. At the end of the operation, the operation site will be checked and hemostasis will be provided. The operator will record the operation in the source documentation. 2 ± 1 days later, a postoperative CT scan will be taken. A follow-up visit will be due 14 ± 2 weeks later, after the osseointegration period.
  Arms: FULL GUIDED
Procedure: Guide-pin-assisted Freehand surgery — The regular protocol of the implant surgery will be followed. Before the surgery begins, the patient will be given anesthesia to ensure they are comfortable and pain-free during the procedure. Doctors will go through the digital planning to understand the desired angulation. Then the bony bed will be prepared raising flap from targeted area. Then a guide-pin will be inserted by drilling and through radiographic image the direction will be confirmed. Following the hole of the guide-pin, the implant will be inserted. At the end of the operation, the raised flap will be sewn and hemostasis will be provided. The operator records the operation in the source documentation. 2 ± 1 days later, a postoperative CT scan will be taken. A follow-up visit will be due 14 ± 2 weeks later, after the osseointegration period.
  Arms: FREE HAND (GUIDE-PIN-assisted)

SUMMARY:
This is a randomized controlled study that aims to compare the accuracy between full-guided with guide-pin-assisted free-hand dental implant surgeries. The basis of evaluation in each case is the comparison of the preoperative digital plan with the actual postoperative status.

DETAILED DESCRIPTION:
Dental implant surgery is a treatment that replaces damaged or missing teeth with artificial teeth that are aesthetically and functionally similar to natural teeth. For a successful implant surgery, it is necessary to use digital planning software in conjunction with a cone-beam CT scan and a custom-made 3D-printed surgical guide. In developing countries like Bangladesh, surgical guide-assisted dental implant surgery is absent. Doctors attend implant surgeries relying on their visual assessment from x-ray images or CBCT data. They need to cut the outer soft tissue, expose the bone, and use a guide pin to confirm the direction and location. Then they perform implant surgery following the hole created by the guide pin, similar to free-hand surgery. But the overall procedure is still highly invasive and has low accuracy.

Free-hand implant surgeries are still in practice everywhere. The application of a guide pin has been observed in some places to enhance the situation. A guide pin helps an operator recognize the position and angle of an alveolar bone when forming an implantation hole in the alveolar bone to insert an implant into the alveolar bone. Doctors insert a guide pin to the implant site with minimal incision and then confirm the desired direction and location with a radiographic image. However, we need a proper clinical evaluation to compare fully-guided surgeries to guide-pin-assisted surgeries to understand the accuracy of both processes.

The accuracy of the pre-planned 3D-printed surgical guide is well established. Introducing dental software and guided surgery has already achieved higher acceptance in implant surgery. Several patients from several privileged parts of the world benefit from surgical guides. But the usual design convention includes intraoral scanner data with CBCT. However, intraoral scanners are still unavailable in many dental hospitals. The study is designed to address the precision of dental implant surgeries worldwide, especially where the intraoral scanner is not present. In our research, we will focus on partially edentulous patients. And our design procedure will not be dependent on intra-oral scanner data. As partially edentulous patients are higher in number and CBCT machines readily available in hospitals, this study can open up a way to address the scarcity of intra-oral scanner data to avail a large number of implant patients with an effective guide. The success rate of this study will encourage us not only to prioritize guided surgeries over free-hand practices or guide-pin-assisted surgeries but also to significantly impact the execution of implant surgeries in developing countries.

ELIGIBILITY:
Inclusion Criteria:

* Patients of age between 18 to 75 and of any gender
* Patient fit for implantation (satisfactory soft and hard tissue conditions and occlusion)
* Partially edentulous patient

Exclusion Criteria:

* Patient with pregnancy
* Patient with uncontrolled diabetes mellitus.
* Patient who needed dentoalveolar or associated soft tissue reconstruction procedure
* Patient taking bisphosphonate or have any history of systemic or local bone disease
* Recent extracted sites
* Patients with a history of smoking, alcoholism
* Patient with a history of head-neck radiation
* Patient with associated periapical pathology or history of parafunctional habit
* Patient needs bone grafting.
* Known HIV, Hepatitis B, or Hepatitis C infection.
* Limited mouth opening, which, in the examiner's opinion, would risk the success of the intervention
* Local infection
* Known allergy to any component of the implant or the implant guide

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2023-08-23 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Angular deviation | 3 months
  The angle formed by the primary axis of the proposed digital implant and the actual implant as put, stated in degrees.

SECONDARY OUTCOMES:
Apical deviation | 3 months
  The deviation of the implant's apical point from the anticipated apical position in three dimensions, measured in millimeters.
Coronal deviation | 3 months
  The deviation of the implant's coronal point from the anticipated coronal position in three dimensions, measured in millimeters.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Md Al-Amin Sarkar, BDS, FCPS (Prosthodontics), Principal Investigator — Dhaka Dental College Hospital
Locations (1):
- Dhaka Dental College and Hospital, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Albrektsson T, Dahl E, Enbom L, Engevall S, Engquist B, Eriksson AR, Feldmann G, Freiberg N, Glantz PO, Kjellman O, et al. Osseointegrated oral implants. A Swedish multicenter study of 8139 consecutively inserted Nobelpharma implants. J Periodontol. 1988 May;59(5):287-96. doi: 10.1902/jop.1988.59.5.287. PMID 3290429
- [Background] Bacchetti P, Leung JM. Sample size calculations in clinical research. Anesthesiology. 2002 Oct;97(4):1028-9; author reply 1029-32. doi: 10.1097/00000542-200210000-00050. No abstract available. PMID 12357184
- [Background] Cassetta M, Stefanelli LV, Giansanti M, Di Mambro A, Calasso S. Depth deviation and occurrence of early surgical complications or unexpected events using a single stereolithographic surgi-guide. Int J Oral Maxillofac Surg. 2011 Dec;40(12):1377-87. doi: 10.1016/j.ijom.2011.09.009. Epub 2011 Oct 15. PMID 22001378
- [Background] Coravos A, Goldsack JC, Karlin DR, Nebeker C, Perakslis E, Zimmerman N, Erb MK. Digital Medicine: A Primer on Measurement. Digit Biomark. 2019 May 9;3(2):31-71. doi: 10.1159/000500413. eCollection 2019 May-Aug. PMID 32095767
- [Background] Geng W, Liu C, Su Y, Li J, Zhou Y. Accuracy of different types of computer-aided design/computer-aided manufacturing surgical guides for dental implant placement. Int J Clin Exp Med. 2015 Jun 15;8(6):8442-9. eCollection 2015. PMID 26309497
- [Background] Israelson H, Plemons JM, Watkins P, Sory C. Barium-coated surgical stents and computer-assisted tomography in the preoperative assessment of dental implant patients. Int J Periodontics Restorative Dent. 1992;12(1):52-61. PMID 1526711
- [Background] Jacobs R, Adriansens A, Verstreken K, Suetens P, van Steenberghe D. Predictability of a three-dimensional planning system for oral implant surgery. Dentomaxillofac Radiol. 1999 Mar;28(2):105-11. doi: 10.1038/sj/dmfr/4600419. PMID 10522199
- [Background] Jacobs R, Adriansens A, Naert I, Quirynen M, Hermans R, Van Steenberghe D. Predictability of reformatted computed tomography for pre-operative planning of endosseous implants. Dentomaxillofac Radiol. 1999 Jan;28(1):37-41. doi: 10.1038/sj.dmfr.4600403. PMID 10202477
- [Background] Kernen F, Benic GI, Payer M, Schar A, Muller-Gerbl M, Filippi A, Kuhl S. Accuracy of Three-Dimensional Printed Templates for Guided Implant Placement Based on Matching a Surface Scan with CBCT. Clin Implant Dent Relat Res. 2016 Aug;18(4):762-8. doi: 10.1111/cid.12348. Epub 2015 Apr 28. PMID 25923363
- [Background] Kiatkroekkrai P, Takolpuckdee C, Subbalekha K, Mattheos N, Pimkhaokham A. Accuracy of implant position when placed using static computer-assisted implant surgical guides manufactured with two different optical scanning techniques: a randomized clinical trial. Int J Oral Maxillofac Surg. 2020 Mar;49(3):377-383. doi: 10.1016/j.ijom.2019.08.019. Epub 2019 Sep 20. PMID 31543382
- [Background] Lin CC, Ishikawa M, Maida T, Cheng HC, Ou KL, Nezu T, Endo K. Stereolithographic Surgical Guide with a Combination of Tooth and Bone Support: Accuracy of Guided Implant Surgery in Distal Extension Situation. J Clin Med. 2020 Mar 5;9(3):709. doi: 10.3390/jcm9030709. PMID 32151043
- [Background] Schneider D, Marquardt P, Zwahlen M, Jung RE. A systematic review on the accuracy and the clinical outcome of computer-guided template-based implant dentistry. Clin Oral Implants Res. 2009 Sep;20 Suppl 4:73-86. doi: 10.1111/j.1600-0501.2009.01788.x. PMID 19663953
- [Background] Verstreken K, Van Cleynenbreugel J, Martens K, Marchal G, van Steenberghe D, Suetens P. An image-guided planning system for endosseous oral implants. IEEE Trans Med Imaging. 1998 Oct;17(5):842-52. doi: 10.1109/42.736056. PMID 9874310
- [Background] Younes F, Cosyn J, De Bruyckere T, Cleymaet R, Bouckaert E, Eghbali A. A randomized controlled study on the accuracy of free-handed, pilot-drill guided and fully guided implant surgery in partially edentulous patients. J Clin Periodontol. 2018 Jun;45(6):721-732. doi: 10.1111/jcpe.12897. Epub 2018 May 10. PMID 29608793
- [Background] D'haese J, Van De Velde T, Komiyama A, Hultin M, De Bruyn H. Accuracy and complications using computer-designed stereolithographic surgical guides for oral rehabilitation by means of dental implants: a review of the literature. Clin Implant Dent Relat Res. 2012 Jun;14(3):321-35. doi: 10.1111/j.1708-8208.2010.00275.x. Epub 2010 May 11. PMID 20491822
- [Background] Wang X, Ji X. Sample Size Estimation in Clinical Research: From Randomized Controlled Trials to Observational Studies. Chest. 2020 Jul;158(1S):S12-S20. doi: 10.1016/j.chest.2020.03.010. PMID 32658647